CLINICAL TRIAL: NCT01682564
Title: Open Label, Randomized, Active Drug Comparative, Parallel Group, Multi-center, Phase IV Study to Compare and Evaluate the Efficacy and Safety of Candemore Tab and Atacand Tab.
Brief Title: To Evaluate the Efficacy and Safety on Blood Pressure In Patients With Hypertension Diagnosed Congestive Heart Failure
Acronym: CANTABILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: m106CHF11E
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Hypertension; Congestive Heart Failure
Keywords: Candemore; Atacand; Candesartan cilexetil; Primary Hypertension; Congestive Hypertension
MeSH Terms: conditions — Hypertension; Heart Failure; Essential Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candemore tablet (Experimental): Candemore tablet
  * Initial dose : 4mg/day if SBP<140mmHg and/or DBP<90mmHg, 8mg/day if SBP≥140mmHg and DBP≥90mmHg
  * dose escalation : double dose if SBP≥100mmHg and DBP>60mmHg (maximum dose 16mg/day)
  Interventions: Drug: Candemore tablet
- Atacand tablet (Active Comparator): Atacand tablet
  * Initial dose : 4mg/day if SBP<140mmHg and/or DBP<90mmHg, 8mg/day if SBP≥140mmHg and DBP≥90mmHg
  * dose escalation : double dose if SBP≥100mmHg and DBP>60mmHg (maximum dose 16mg/day)
  Interventions: Drug: Atacand tablet

INTERVENTIONS:
Drug: Candemore tablet — * Initial dose : 4mg/day if SBP<140mmHg and/or DBP<90mmHg, 8mg/day if SBP≥140mmHg and DBP≥90mmHg
  * dose escalation : double dose if SBP≥100mmHg and DBP>60mmHg (maximum dose 16mg/day)
  Arms: Candemore tablet
Drug: Atacand tablet — * Initial dose : 4mg/day if SBP<140mmHg and/or DBP<90mmHg, 8mg/day if SBP≥140mmHg and DBP≥90mmHg
  * dose escalation : double dose if SBP≥100mmHg and DBP>60mmHg (maximum dose 16mg/day)
  Arms: Atacand tablet

SUMMARY:
To compare and evaluate the efficacy and safety of Candemore tab. versus Atacand tab. on blood pressure in patients with hypertension diagnosed congestive heart failure

DETAILED DESCRIPTION:
This is an open label, randomized, active drug comparative, Parallel group, Multi-center, phase IV study. Patients receive candemore tablet or atacand tablet. Initial dose is 4mg/day or 8mg/day. Every 2 weeks, patients take double dose if patients blood pressure is measured SBP ≥ 100mmHg and DBP > 60mmHg. Maximum dose is 16mg/day.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to provide written informed consent
* age 20 years or older
* patient with congestive heart failure, taking treatment medicine and NYHA grade II~III
* patient with hypertension, taking treatment medicine or SBP ≥ 140mmHg or DBP ≥ 90mmHg at the screening visit

Exclusion Criteria:

* Known or suspected secondary hypertension(ex. aortic coactation, primary hyperaldosteronism, renal artery stenosis, pheochromocytoma, cushing syndrome, polycystic renal disease)
* blood creatinine level ≥ 2.5mg/dl
* blood potassium level > 5.5mEq/L
* blood SGOT, SGPT level ≥ maximum normal range X3 or patient with sever hepatic dysfunction, cholestasis
* pregnant or breast-feeding
* premenopausal women not using adequate contraception
* patient has history about hypersensitivity or taboo of investigational product
* patient with lactose intolerance or Lapp lactase deficiency or glucode-galactose malabsorption
* administration of other study drugs within 1 month prior to screening
* history of ischemic heart disease(ex. angina pectoris, myocardial infarction) within the last 3 months
* in investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mean sitting Systolic Blood Pressure | After 12 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure | After 12 weeks of treatment
echocardiography | After 12 weeks of treatment
  Left Ventricle Volume, Left Ventricle Ejection Fraction, E/E' ration, Peak TR velocity
Blood Creatinine and Potssium level | After 4 and 12 weeks of treatment
NYHA class | After 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: KeeSik Kim, M.D Ph.D, Principal Investigator — Daegu Catholic University Medical Center
Locations (14):
- South Korea (14):
  - Inje university pusan hospital, Busan, Busanjin-gu Gaegum-dong
  - Gyeongsang national university hospital, Jinju, Chiram-dong
  - Daegu fatima hospital, Daegu, Dong-gu Sinam-dong
  - Daedong hospital, Busan, Dongnae-gu Myeongnyun-dong
  - Inje university haeundae paik hospital, Busan, Haeundae-gu Heaundae-ro 875
  - Maryknoll medical center, Busan, Jung-gu Daecheong-dong
  - Keimyung university dongsan medical center, Daegu, Jung-gu Dongsan-dong
  - Kyungpook national university hospital, Daegu, Jung-gu Samdeok-dong
  - Samsung changwon hospital, Changwon, Masanhoiwon-gu Hapseong-dong 50
  - Yeungnam university medical center, Daegu, Nam-gu Daemyeong-dong
  - Daegu catholic univ. medical center, Daegu, Nam-gu Daemyung-dong
  - Kosin university gospel hospital, Busan, Seo-gu Amnam-dong
  - Dong-A university medical center, Busan, Seo-gu Dongdaesin-dong
  - Dongguk university gyeongju hospital, Gyeongju, Seokjang-dong